CLINICAL TRIAL: NCT05327218
Title: Effectiveness and Safety of Preoperative Magnetic Detection of Non-palpable Breast Lesions
Acronym: MAGREES
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MAGREES
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Diseases; Breast Cancer
MeSH Terms: conditions — Breast Diseases; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common cancer in women and also has the highest death rate. In 2018, 58,500 new cases were diagnosed in metropolitan France. It affects, in 8 out of 10 cases, women aged 50 and over. Nevertheless, thanks to early detection and improved therapeutic techniques, its mortality rate has continued to decrease each year (a decrease of 1.6% per year was recorded between 2010 and 2018), which allows it to maintain its status as a cancer with a good prognosis. Furthermore, net survival is 87% at 5 years and 76% at 10 years. The median age of death is 74 years. Organized screening was initiated in France in 1990 and generalized in 2004, while maintaining a specific management according to the personal risk of each patient. It consists of a mammogram, plus or minus an ultrasound, every two years from the age of 50. The mammogram is reviewed by two different radiologists. In case of abnormality, a biopsy is performed.

Breast lesions are separated into two nosological entities: palpable tumors, often diagnosed on clinical examination (or autopalpation) and confirmed on mammography, and non-palpable tumors detected during mammographic and/or ultrasound screening.

Thanks to the generalization of screening, the detection of subclinical lesions requiring surgery represents more than half of the breast surgeries and the challenge of their surgical management lies in a precise preoperative location to allow a complete removal, while limiting the sacrifice of healthy glandular tissue. The metallic location technique is currently the reference technique for the preoperative location of these lesions.

For all these reasons, new techniques of preoperative tracking have been developed.

Magnetic tracking (MR) appears to be a simple, non-radioactive and non-aggressive technique to use and organize. MR takes the form of a 1x5mm paramagnetic clip made of iron oxide visible on ultrasound and mammography and is detected by a SentiMag probe. The MR began to be used in France in 2017. It is placed in contact with the lesion under ultrasound guidance. It has the advantage that it can be placed up to 30 days before surgery and has less risk of complication. This MR contains iron particles and is 5mm long. It is pre-loaded in a sterile 18 G needle closed with a wax tip. It is deployed under mammographic and/or ultrasound guidance. The Sentimag probe is used to detect MR in a multidirectional way at 360°, with an audio and visual estimation of the distance. It generates an alternating magnetic field that magnetizes the iron in the MR.

All of these surgical procedures can be performed as outpatient surgery, which corresponds to a hospitalization of less than 12 hours without overnight accommodation, meaning that each patient is admitted and discharged on the same day as her procedure. Outpatient surgery represented 36% of all surgeries in France in 2018. The objective of the HAS is to achieve a majority ambulatory practice of 70% by 2022. This type of surgery has advantages for the patient, by making her journey safer: reduction in the risk of nosocomial infection, thromboembolic risk and anxiety linked to hospitalization for the patient and her family. It also has an important socio-economic advantage by reducing hospitalization costs and the number of hospital beds required. It improves the working conditions of the staff by reducing the workload and night shifts. It has also enabled a clear improvement in the optimization and efficiency of the organization of resources in the surgical technical platforms. The role of the MR is particularly well suited to this new organization.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with non-palpable benign, atypical or cancerous lesions
* Preoperative biopsy
* Requiring surgical excision
* French speaking patient

Exclusion Criteria:

* Palpable breast lesion
* Contraindication to the installation of a magnetic tracer
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient opposing the use of his data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were or are referred for surgical management of non-palpable breast lesions between May 15, 2018 and December 21, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of magnetic tracking | Day 1
  This outcome corresponds to the number of patients with complete removal of the target lesion.

SECONDARY OUTCOMES:
Safety of magnetic tracking | Day 1
  This outcome corresponds to the occurrence of complications related to the placement of the metallic or magnetic marker.

CONTACTS AND LOCATIONS:
Overall Officials: Severine ALRAN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Broeders M, Moss S, Nystrom L, Njor S, Jonsson H, Paap E, Massat N, Duffy S, Lynge E, Paci E; EUROSCREEN Working Group. The impact of mammographic screening on breast cancer mortality in Europe: a review of observational studies. J Med Screen. 2012;19 Suppl 1:14-25. doi: 10.1258/jms.2012.012078. PMID 22972807
- [Background] Shapiro S. Periodic screening for breast cancer: the HIP Randomized Controlled Trial. Health Insurance Plan. J Natl Cancer Inst Monogr. 1997;(22):27-30. doi: 10.1093/jncimono/1997.22.27. PMID 9709271
- [Background] Chagpar AB, Garcia-Cantu C, Howard-McNatt MM, Gass JS, Levine EA, Chiba A, Lum S, Martinez R, Brown E, Dupont E; SHAVE2 authors. Does Localization Technique Matter for Non-palpable Breast Cancers? Am Surg. 2022 Dec;88(12):2871-2876. doi: 10.1177/00031348211011135. Epub 2021 Apr 15. PMID 33856948
- [Background] Hall FM, Frank HA. Preoperative localization of nonpalpable breast lesions. AJR Am J Roentgenol. 1979 Jan;132(1):101-5. doi: 10.2214/ajr.132.1.101. PMID 103383
- [Background] Frank HA, Hall FM, Steer ML. Preoperative localization of nonpalpable breast lesions demonstrated by mammography. N Engl J Med. 1976 Jul 29;295(5):259-60. doi: 10.1056/NEJM197607292950506. No abstract available. PMID 934190
- [Background] Norman C, Lafaurie G, Uhercik M, Kasem A, Sinha P. Novel wire-free techniques for localization of impalpable breast lesions-A review of current options. Breast J. 2021 Feb;27(2):141-148. doi: 10.1111/tbj.14146. Epub 2020 Dec 27. PMID 33368757
- [Background] Jeffries DO, Dossett LA, Jorns JM. Localization for Breast Surgery: The Next Generation. Arch Pathol Lab Med. 2017 Oct;141(10):1324-1329. doi: 10.5858/arpa.2017-0214-RA. PMID 28968154
- [Background] Pieszko K, Wichtowski M, Cieciorowski M, Jamont R, Murawa D. Evaluation of the nonradioactive inducible magnetic seed system Magseed for preoperative localization of nonpalpable breast lesions - initial clinical experience. Contemp Oncol (Pozn). 2020;24(1):51-54. doi: 10.5114/wo.2020.93677. Epub 2020 Mar 13. PMID 32514238
- See also: Related Info — https://www.e-cancer.fr/Professionnels-de-sante/Les-chiffres-du-cancer-en-France/Epidemiologie-des-cancers/Les-cancers-les-plus-frequents/Cancer-du-sein
- See also: Cancer du sein (II). Procédures diagnostiques et thérapeutiques — https://www.em-consulte.com/article/225924/cancer-du-sein-ii-procedures-diagnostiques-et-ther